CLINICAL TRIAL: NCT07156123
Title: Analysis of Safety and Efficacy of Long-term Treatment With PD Catheters
Brief Title: PD Catheter Data Collection
Acronym: Catheter
Status: Not yet recruiting | Type: Observational
Sponsor: Fresenius Medical Care Deutschland GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: PD-Cathether-01-INT
Record Dates: First submitted 2025-05-21; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Renal Insufficiency / Therapy
Keywords: Peritoneal dialysis; Renal replacement therapy; Ultrafiltration; Catheter
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PD treatment: Include all the patients treated with peritoneal dialysis (PD or APD) using the PD catheter as described and who who will begin PD, or patients who began PD within the last 1.5 years before start of the study

SUMMARY:
Peritoneal Dialysis (PD) is a Renal Replacement Therapy for patients with renal insufficiency that has been used more frequently in recent years. In PD treatment, catheter are used to provide access to the peritoneal cavity, allowing the dialysate to be introduced and removed from the abdomen. The aim of this study is to evaluate the safety and efficacy of long-term treatment with PD catheters (developed by Fresenius Medical Care (FME)) in adult and paediatric patients treated with CAPD or APD. Safety and performance parameters of the catheters will be analyzed, as well as data on PD treatment outcome, such as Peritoneal Clearance and Peritoneal Ultrafiltration.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent for study participation and data submission (by the patient or legal representative for patients under 18) along with investigator/authorized physician signature.
* Patients under 18 who have received age- and maturity-appropriate information per Article 63(2) MDR from trained investigators or team members; minors capable of understanding must also sign the informed consent.
* The investigator must respect the decision of any minor, capable of understanding the information as per Article 63(2) MDR, to decline participation or withdraw from the clinical investigation at any time.
* Ability to understand the nature and requirements of the study.
* Patients with indication for renal replacement therapy, specifically PD (CAPD or APD)
* Patients who began PD using FME catheters within the last 18 months and are either prevalent in PD at study initiation or have switched to HD or undergone transplantation and can consent to data use.
* Incident patients who will begin PD using FME catheters.

Exclusion Criteria:

* Patient or legal representative is not able to give informed consent according to European Medical Device Regulation and corresponding national regulations,
* Previous participation in the same study.
* Life expectancy < 3 months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the patients treated with peritoneal dialysis (PD or APD) using the PD catheter as described and who who will begin PD, or patients who began PD within the last 1.5 years before start of the study
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Safety variables | Every 6 months (± 2 months, as per centre practice)
  Catheter related infections (e.g. peritonitis, tunnel infections, exit site infection)
Safety variables | Every 6 months (± 2 months, as per centre practice)
  Non-infectious complications
Safety variables | Every 6 months (± 2 months, as per centre practice)
  Biocompatibility (allergic reaction)
Safety variables | Every 6 months (± 2 months, as per centre practice)
  Identify new emerging risks
Safety variables | Every 6 months (± 2 months, as per centre practice)
  Monitor side effects
Safety variables | Every 6 months (± 2 months, as per centre practice)
  Catheter removal

SECONDARY OUTCOMES:
Performance variables | very 6 months (± 2 months, as per centre practice)
  Catheter patency
Performance variables | very 6 months (± 2 months, as per centre practice)
  Non-infectious complication
Outcome variables | very 6 months (± 2 months, as per centre practice)
  Peritoneal clearance
Outcome variables | very 6 months (± 2 months, as per centre practice)
  Peritoneal UF
Outcome variables | very 6 months (± 2 months, as per centre practice)
  Mechanical complications
Outcome variables | very 6 months (± 2 months, as per centre practice)
  Therapy tolerability.